CLINICAL TRIAL: NCT02875301
Title: Investigating Gains in Neurocognition in an Intervention Trial of Exercise
Acronym: IGNITE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kirk Erickson, PhD, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY19070071; R01AG053952 (NIH); R01AG060050 (NIH)
Record Dates: First submitted 2016-08-12; First posted 2016-08-23 (Estimated); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Healthy; Cognitive Function 1, Social
Keywords: Exercise; Brain Health; Dose Response; Cognition
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Study participants will be randomly assigned to one of three exercise intervention arms.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 150 Minutes Week (Experimental): Participants engage in supervised 12 month moderate intensity aerobic exercise intervention with goal of maintaining 150 minutes of exercise per week.
  Interventions: Behavioral: 150 Minutes Week
- 225 Minutes Week (Experimental): Participants engage in supervised 12 month moderate intensity aerobic exercise intervention with goal of maintaining 225 minutes of exercise per week.
  Interventions: Behavioral: 225 Minutes Week
- Stretch and Tone (Active Comparator): Participants engage in supervised 12 month non-cardiorespiratory activity intervention. This group has focus on improving balance, flexibility, and strength.
  Interventions: Behavioral: Stretch and Tone

INTERVENTIONS:
Behavioral: 150 Minutes Week — This group will complete aerobic based exercise 150 minutes per week. Participants will obtain minutes through supervised on site exercise and home based exercise. An exercise duration of 30 minutes will be achieved by the forth week of the program and be maintained for the duration of the intervention. Heart rate will be monitored to ensure proper intensity levels. Participants will also be instructed to exercise at home for 30 minutes for two other days of the week at a similar intensity. The prescribed intensity will be 50-60% of the maximum heart rate reserve for weeks one to six and 60-75% for the remainder of the program. Participants in the walking conditions will wear heart rate monitors and be encouraged to walk within their target heart rate zone. During the Covid-19 pandemic shutdown, all intervention exercise was been shifted to home based.
  Arms: 150 Minutes Week
Behavioral: 225 Minutes Week — This group will complete aerobic based exercise 225 minutes per week. Participants will obtain minutes through supervised on site exercise and home base exercise. A walking duration of 45 minutes will be achieved by the seventh week of the program. This will be maintained for the duration of the intervention and heart rate will be monitored to ensure proper intensity levels. Participants will be instructed to exercise at home for 45 minutes for two other days of the week at a similar intensity. The prescribed intensity will be 50-60% of the maximum heart rate reserve for weeks one to six and 60-75% for the remainder of the program. Participants in the walking conditions will wear heart rate monitors and be encouraged to walk within their target heart rate zone. During the Covid-19 pandemic shutdown, all intervention exercise has been shifted to home based.
  Arms: 225 Minutes Week
Behavioral: Stretch and Tone — The control condition will focus on improving balance, flexibility, and strength. This group will obtain 150 minutes per week via in person sessions, zoom sessions and home based stretching. Resistance bands, balance disks, yoga blocks, and exercise mats will be used to engage in non-cardiorespiratory activities. These are progressive in nature and include modifications to accommodate injuries, physical difficulties, etc. A new set of similar, yet slightly more challenging activities will be introduced every four weeks. During the first two weeks, participants are introduced to the new activities, and, during the second two weeks, they are encouraged to increase intensity by using more weight or more repetitions. During the current Covid-19 pandemic, all intervention exercise has been shifted to home based.
  Arms: Stretch and Tone

SUMMARY:
This randomized control trial will examine whether a 12 month monitored exercise intervention improves brain health in cognitively normal older adults. This trial will also address several important unanswered questions: (1) Are the recommended public health guidelines of 150 minutes/week of exercise sufficient for improving cognitive performance? (2) Does exercise influence brain structure and/or function? (3) Is there a dose-response effect of exercise on the above variables such that greater amounts of exercise brings about greater benefits in cognitive and brain health? (4) What are the mechanisms by which exercise influences brain health? and (5) What factors attenuate or magnify the effects of exercise on brain and cognitive health and contribute to the individual variability in intervention outcomes?

DETAILED DESCRIPTION:
The investigators are conducting a 12-month, multi-site, randomized dose-response exercise trial (i.e., brisk walking) in 639 cognitively normal adults between 65-80 years of age. Participants will be randomized to a (a) moderate intensity aerobic exercise condition at the public health recommended dose of 150 minutes/week (N=213), (b) a moderate intensity exercise condition at 225 minutes/week (N=213), or (c) a light intensity stretching-and-toning control condition for 150 minutes per week (N=213). Participants will meet 3 days/week for site-based exercise and do home-based activity on two more days of the week for 12 months. A comprehensive state-of-the-science battery of cognitive, MRI, amyloid imaging, physiological biomarkers, cardiorespiratory fitness, physical function, and quality of life measures will be assessed at baseline and after completion of the intervention.

Due to Covid-19 pandemic, the exercise intervention was moved to fully home based during the months of March 2020 through August 2020. During this time, study participants were mailed wrist based heart rate monitors to track intensity. Exercise videos were developed and released to study participants to enhance adherence to the prescribed volume of exercise. Study participants were contacted weekly to obtain weekly exercise volume, mode and intensity. From August 2020 to end of the trial, participants will have flexibility to complete randomized goal of exercise. The study recommends three supervised sessions per week but will work with study participants who feel unsafe exercising in one of the study locations.

The outcome measures to be collected during March 2020 and July 2020 were delayed in those subjects had original intervention end date during this time. For these study participants, many signed a study consent extension and continued the intervention until study sites were allowed to re-open after careful planning and approved mitigation plans at each respective university. Once approved to re-open, participants were scheduled for their post assessment outcome collection.

Specific Aims include:

1. Cognitive Enhancement: Using a comprehensive neuropsychological battery and the NIH Toolbox, the investigators will test (a) whether a 12-month moderate intensity exercise intervention improves cognitive performance in older adults and (b) whether the improvements occur in a dose-dependent manner. Hypothesis: PA will enhance cognitive performance non-uniformly with the greatest effects occurring for executive and declarative memory functions. The investigators also predict that these improvements will follow a dose-dependent trajectory with 225 minutes/week of PA demonstrating greater improvements than 150 minutes/week of PA.
2. Brain Augmentation: The investigators will test (a) whether a 12-month PA intervention augments MRI markers of brain health and (b) whether changes happen in a dose-dependent manner. Hypothesis: PA will most profoundly influence the volume, microstructural white matter integrity, cerebral blood flow, and connectivity of regions supporting declarative memory (e.g., hippocampus) and executive function (e.g., prefrontal cortex; PFC). Further, the investigators predict that 225 minutes/week will result in greater effects than 150 minutes/week. The investigators predict that these changes in brain outcomes will mediate the cognitive improvements in Aim 1.
3. Biomediators: The investigators will test the hypothesis that cardiometabolic, inflammatory, and neurotrophic changes mediate improvements in brain and cognition. Hypothesis: (1) decreases in pro-inflammatory cytokines, (2) decreases in central adiposity, arterial stiffness, and insulin resistance, and (3) increases in brain-derived neurotrophic factor (BDNF) levels will statistically mediate changes in cognitive performance (Aim 1) and brain health (Aim 2), and that the strength of this mediating relationship might vary as a function of certain apriori moderating variables of interest
4. Moderators: To examine subgroups (i.e., individual differences) that attenuate or magnify the effect of the intervention on cognitive, brain, and physiological systems to better understand the factors that predict 'responders' versus 'non-responders' to the intervention. The investigators will examine three categories of variables: (1) demographic (e.g., age) (2) genetic (e.g., APOE), and (3) baseline Aβ burden. Hypothesis: The favorable effects of PA on brain and cognition will be greatest for older individuals with greater Aβ burden, and in those with a genetic susceptibility for accelerated cognitive decline.
5. Amyloid Diminution: We will test (a) assess Amyloid deposition changes in response to physical activity and (b) whether changes occur in a dose-dependent manner and (c) examine baseline Amyloid as a moderator of intervention effects and (d) examine changes in Amyloid as a mediator of changes in brain and cognition. Hypothesis: We predict that Aβ burden will be attenuated over the course of the intervention for the aerobic exercise groups compared to control group. Further, we predict that 225 minutes/week of aerobic exercise will result in a greater effect on Aβ than 150 minutes/week
6. Exploratory Aims: The investigators will explore (a) whether baseline brain health metrics predict adherence and compliance to 12-months of PA, and (b) the utility of multi-modal brain imaging analytical approaches to more comprehensively understand the effects of PA on the aging brain.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 65 - 80 yrs
* Ambulatory without pain or the assistance of walking devices
* Able to speak and read English
* Exercise level of <60 minutes per week (less than 20 minutes / 3 days week)
* Medical clearance by PCP
* Living in community for duration of the study
* Reliable means of transportation
* No diagnosis of a neurological disease
* Eligible to undergo MRI

Exclusion Criteria:

* Current diagnosis of a DSM-V Axis I or II disorder including Major Depression
* History of major psychiatric illness including schizophrenia (not including general anxiety disorder or depression)
* Current treatment for cancer - except non-melanoma skin
* Neurological condition (MS, Parkinson's, Dementia, MCI) or brain injury (traumatic or Stroke)
* Type I Diabetes or insulin-dependent diabetes
* Current alcohol or substance abuse
* Current treatment for congestive heart failure, angina, uncontrolled arrhythmia, DVT or other cardiovascular event
* Myocardial infarction, coronary artery bypass grafting, angioplasty or other cardiac condition in the past year
* Regular use of an assisted walking device
* Presence of metal implants (pacemaker, stents) that would be MR ineligible
* Claustrophobia
* Color Blindness
* Not fluent in English
* Not medically cleared by PCP
* Engaging in >60 minutes of moderate intensity physical activity (more than 20 minutes day / 3 days per week)
* Traveling consecutively for 3 weeks or greater during the study

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 648 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Function | Baseline and 12 months
  Investigators are assessing change in cognitive function from baseline to 12 months. A comprehensive neuropsychological battery will be used that assesses 5 domains of cognitive function (Working Memory, Processing Speed, Episodic Memory, Attentional Control, and Visuospatial Function). We will perform a confirmatory factor analysis on the cognitive data and determine whether the exercise intervention influences performance as measured by these factors. There is no min and max values. These are generated from a confirmatory factor analysis that normalizes the scores around 0 (being the mean). As such, positive values reflect better performance and negative values reflect poorer cognitive performance. Since the scores are standardized we can calculate the changes in standard deviations - e.g., a shift of 0.5 would be an improvement of ½ standard deviation in performance based on the sample average.

SECONDARY OUTCOMES:
Change in brain morphology (Volume) | Baseline and 12 months
  MRI will be used to measure average hippocampal volume and determine changes in volume over the course of the intervention.

OTHER OUTCOMES:
Change in white matter lesions | Baseline and 12 months
  MRI will be used to measure the number of white matter lesions before and after the intervention.
Change in hippocampal subfield volumes | Baseline and 12 months
  MRI will be used to measure volumetric changes in hippocampal subfields.
Change in cortical thickness | Baseline and 12 months
  MRI will be used to measure average cortical thickness over the course of the intervention.
Change in cerebral blood flow | Baseline and 12 months
  MRI will be used to measure changes in cerebral blood flow. Total cerebral blood flow changes over the course of the intervention will be evaluated.
Change in resting state brain activity | Baseline and 12 months
  MRI will be used to measure changes in resting state brain function. We will examine whether the intervention alters resting state connectivity metrics.
Change in white matter diffusion properties | Baseline and 12 months
  MRI will be used to measure changes in white matter microstructure in relation to the intervention.
Change in task-evoked relational memory brain activity | Baseline and 12 months
  MRI will be used to measure changes in encoding and retrieval during a relational memory task.
Change in task-evoked working memory brain activity | Baseline and 12 months
  MRI will be used to measure changes in brain activity task-evoked patterns using an N-back working memory task.
APOE Status | Baseline
  The APOE e4 carrier status increases risk for Alzheimer's disease. We will be examining whether any outcomes are moderated by carriage of the APOE e4 allele.
Change in blood levels of brain-derived neurotrophic factor (BDNF) | Baseline, 6 Months, and 12 Months
  BDNF helps regulate synaptic plasticity, which is important for learning and memory and might change in response to exercise. We will be evaluating whether changes in BDNF mediate changes in brain or cognitive outcomes.
Change in blood levels of inflammatory cytokines - TNF-Alpha | Baseline, 6 Months, and 12 Months
  Exercise might alter cognitive and brain processes by influencing markers of systemic inflammation including TNF-alpha. We will examine whether exercise alters this marker and whether it relates to changes in neurocognitive outcomes.
Change in blood levels of inflammatory cytokines - IL-6 | Baseline, 6 Months, and 12 Months
  Exercise might alter cognitive and brain processes by influencing markers of systemic inflammation including IL-6. We will examine whether exercise alters this marker and whether it relates to changes in neurocognitive outcomes.
Change in blood levels of insulin-like growth factor | Baseline, 6 Months, and 12 Months
  IGF-1 is responsive to exercise and might influence brain and cognitive outcomes in late adulthood. We will examine whether exercise alters this marker and whether it relates to changes in neurocognitive outcomes.
Change in blood levels of vascular endothelial growth factor (VEGF) | Baseline, 6 Months, and 12 Months
  VEGF is responsive to exercise and might influence brain and cognitive outcomes in late adulthood. We will examine whether exercise alters this marker and whether it relates to changes in neurocognitive outcomes.
Change in blood levels of amyloid-beta | Baseline and 12 month
  Amyloid levels measured via blood samples will be examined to determine whether the exercise intervention altered this marker of neuropathology.
Changes in blood levels of p-tau217 | Baseline, 6 months and 12 month
  p-Tau levels measured via blood samples will be examined to determine whether the exercise intervention altered this marker of neuropathology.
Changes in blood levels of p-tau181 | Baseline, 6 months and 12 month
  p-Tau levels measured via blood samples will be examined to determine whether the exercise intervention altered this marker of neuropathology.
Changes in blood levels of p-tau231 | Baseline, 6 months and 12 month
  p-Tau levels measured via blood samples will be examined to determine whether the exercise intervention altered this marker of neuropathology.
Changes in blood levels of glial fibrillary acidic protein (GFAP) | Baseline, 6 months and 12 month
  GFAP levels measured via blood samples will be examined to determine whether the exercise intervention altered this marker of neuropathology.
Changes in blood levels of Neurofilament light | Baseline, 6 months and 12 month
  NFL levels measured via blood samples will be examined to determine whether the exercise intervention altered this marker of neuropathology.
Change in insulin | Baseline, 6 Months, and 12 Months
  We will examine whether changes in markers of insulin resistance (HOMA-IR) change over the course of the intervention and whether these changes mediate neurocognitive outcomes.
Change in glucose | Baseline, 6 Months, and 12 Months
  We will examine whether changes in markers of insulin resistance change over the course of the intervention and whether these changes mediate neurocognitive outcomes.
Change in Cardiorespiratory Fitness | Baseline and 12 Months
  Fitness is assessed by maximal graded exercise testing. Oxygen uptake (VO2) will be measured from expired air samples taken at 15 second intervals until a peak VO2, the highest VO2, is attained at the point of test termination due to symptom limitation and/or volitional exhaustion.
  We will examine whether changes in cardiorespiratory fitness mediates changes to neurocognitive function.
Alzheimer's Disease (AD) PET amyloid | Baseline
  Florbetapir F 18 or Amyvid PET scans are obtained to establish the presence or absence of cerebral amyloidosis. We will examine whether the presence of amyloid moderates the effectiveness of the intervention to influence neurocognitive outcomes.
Change in the trajectory of cognitive function | 6 months
  A subset of the cognitive tests are administered at a midpoint session. These tests will be used to examine trajectories of change on particular cognitive tests. The scores will be generated using similar approaches as for the primary aim but because the tests slightly differ from the baseline and post-intervention assessment, we will have to generate these scores separately. The scores will be normalized so that a 0 represents the mean performance for the sample. Higher values reflect better performance and lower values represent poorer performance
Change in Body Mass Index (BMI) | Baseline and 12 Months
  We will examine whether the intervention altered BMI and whether these changes mediate any changes in behavioral or neurocognitive outcomes.
Change in Visceral Adipose Tissue (VAT) | Baseline and 12 Months
  This will be assessed using a dual-energy x-ray absorptiometer (DXA). The DXA will provide a measure of VAT from a total body scan. We will examine whether the intervention altered VAT levels.
Change in Subcutaneous Adipose Tissue (SAT) | Baseline and 12 Months
  This will be assessed using a dual-energy x-ray absorptiometer (DXA). The DXA will provide a measure of SAT from a total body scan. We will examine whether the intervention altered SAT levels.
Change in Lean mass | Baseline and 12 Months
  This will be assessed using a dual-energy x-ray absorptiometer (DXA). The DXA will provide a measure of lean mass from a total body scan. We will examine whether the intervention altered lean mass levels.
Medical History and Lifestyle habits | Baseline
  Health History assesses medical history and lifestyle habits such as alcohol and tobacco use. We will examine whether any neurocognitive outcomes vary as a function of these health conditions and behaviors.
Medication use | Baseline, 6 months and 12 months
  We will be recording all prescribed and OTC medications that the study participant is currently taking and will examine whether the intervention effects vary as a function of medication use.
Change in quality of life | Baseline, 6 months and 12 months
  We will use the Satisfaction with Life Scale (SWLS) as a global cognitive judgement of study participants life satisfaction. We will examine whether the exercise intervention altered SWLS measures. Total score range is 5 -35 with higher scores equal to greater satisfaction with life.
Change in perceived stress | Baseline, 6 months and 12 months
  The Perceived Stress Scale (PSS) is one of the most widely used psychological instruments for measuring the perception of stress. It measures the degree to which situations in the participants life are gauged as stressful. We will examine whether the exercise intervention modified PSS levels. Score range is 0 - 40 with a higher scores equal to more stress.
Change in health related quality of life (SF-36) | Baseline, 6 months and 12 months
  The SF-36 taps into eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. We will examine whether the exercise intervention modified measures of health related quality of life. Each concept has a score range of 0-100 with higher scores equal to more favorable health traits.
Change in depressive symptoms | Baseline, 6 months and 12 months
  The Hospital Anxiety and Depression Scale (HADS) will be used to measure depressive symptoms. We will examine whether the exercise intervention improved measures of mood and reduced depressive symptoms. Total score range is 0 -21 with lower scores equal to less depressive symptoms.
Change in Mindfulness | Baseline and 12 months
  The MAAS assesses a core characteristic of mindfulness mainly open or receptive awareness of and attention to what is taking place in the present. We will examine whether the exercise intervention altered measures of mindfulness. Score scale runs 15 -90 with higher scores reflecting more mindfulness.
Change in anxiety symptoms | Baseline and 12 months
  The Hospital Anxiety and Depression Scale (HADS) will be used to measure anxiety symptoms. We will examine whether the exercise intervention improved measures of mood and reduced anxiety.
  Total score range 0-21 with lower scores equal to less anxiety symptoms.
SES Composite | Baseline
  Combining information from MacArthur questionnaire to develop Social Economic status of participants. We will examine whether the effectiveness of the intervention varied by SES levels of the participants. The SES composite was generated using a confirmatory factor analysis of various SES indicators - e.g., income, debt, savings, etc. The scores are normalized so that 0 is the average for the sample and higher numbers reflect higher SES and lower numbers indicate lower SES.
Change in Exercise Frequency | Every 2 months starting at baseline until follow-up at 12 months
  Exercise frequency will be measured using Actigraph Link physical activity monitoring device. This device is small and lightweight. It is worn around the non-dominant wrist(touching the skin) for approximately 7 days during all waking and sleeping hours. We will examine whether the intervention altered this measure of daily activity.
Change in Exercise Intensity | Every 2 months starting at baseline until follow-up at 12 months
  Exercise intensity will be measured using the Actigraph Link physical activity monitoring device. This device is small and lightweight. It is worn around the non-dominant wrist (touching the skin) for approximately 7 days during all waking and sleeping hours. We will examine whether the exercise intervention altered amount of time spent in moderate-to-vigorous activities during daily life.
Change in Exercise Duration | Every 2 months starting at baseline until follow-up at 12 months
  Exercise duration will be measured using Actigraph Link physical activity monitoring device. This device is small and lightweight. It is worn around the non-dominant wrist (touching the skin) for approximately 7 days during all waking and sleeping hours.. The duration is measured in minutes. We will examine whether the exercise intervention altered amount of time spent in moderate-to-vigorous activities during daily life.
Change in Reported Fatigue | Baseline, 6 months and 12 months
  Fatigue Symptom Inventory (FSI) is a 14-item self-report measure designed to assess the severity, frequency, and daily pattern of fatigue as well as its perceived interference with quality of life. We will examine whether the exercise intervention impacted perceived daily fatigue. Severity scale score is 0-40 with higher value equal to more severe fatigue. Frequency scale score is 0-21 with higher values meaning more frequent fatigue. Perceived interference scale range is 0-70 with higher values meaning more interference with life.
Change in perceived sleep quality | Baseline and 12 months
  Pittsburgh Sleep Quality Index (PSQI) will be used to assess perceived sleep quality. We will examine whether the exercise intervention alters perceived sleep quality. All components have score range 0-3 with lower number equal to better sleep quality.
Change in optimal time of day | Baseline and 12 months
  The Composite Scale of Morningness assess diurnal preference, sleep times, preferred times for physical and mental activity, and times of subjective alertness. We will examine whether the exercise intervention alters this metric of optimal time of day. scale is 16-86. Score of 70-86 equal morning type, score 59-669 equals moderate morning type, score 42-58 is neither, score 31-41 equals moderate evening type and score 16-30 equal evening type.
Change in subjective cognitive performance | Baseline and 12 months
  Cognitive Function Index (CFI) asks 15 questions in which the participant answers Yes or No to memory items compared to one year prior. We will examine whether the exercise intervention alters subjective cognitive performance. Scoring scale runs 0 - 15 with higher values equal to better cognitive function.
Change in perceived pain | Baseline, 6 months and 12 months
  The McGill Pain Questionnaire is used to evaluate a person's perception of pain. It can be used to monitor the pain over time and to determine the effectiveness of any intervention. We will examine whether the intervention alters perceptions of pain in late adulthood. Score scale runs 0-45 with higher values meaning more pain.
Change in loneliness | Baseline, 6 months and 12 months
  The UCLA Loneliness Scale (UCLA-L) asks subjects to rate, on a scale from 1-4, how often they experience certain feelings. There are 20 feelings listed (e.g. "How often do you feel left out?"). We will examine whether the intervention alters perceptions of loneliness in late adulthood. Scale score is 20-80 with higher values equal to more loneliness.
Change in Fatigue Impact | Baseline and 12 months
  The Brief Fatigue Inventory (BFI) assesses the severity of fatigue and the impact of fatigue on daily functioning. We will examine whether the intervention alters the impact of fatigue on daily function. Higher scores on subscales reflect that participants has that personality. Subscales scores are 8-40 or 9-45.
Prior work history | Baseline
  Work Design Questionnaire (WDQ) gathers information related to the nature and responsibilities of the participant's job. Asks the participant to rate the degree to which he or she agrees (or disagrees) with various questions by "domains" such as job autonomy and complexity, task variety and significance, and cooperative components such as social interactions inside and outside of the organization. We will examine whether changes in cognitive performance varies in relation to the job complexity history.
Change in exercise self-efficacy | Baseline and 12 months
  The investigators will use the Exercise Self-Efficacy Scale (EXSE) to assess belief in the ability to continue exercising three times a week at a moderate intensity for 40 plus minutes a session into the future. We will examine whether this measure predicts long-term adherence outcomes. Score scale runs 0 - 100 with higher values = higher confidence to continue to exercise (3X's week for 40 + minutes) in the future 8 weeks
Change in lower extremity performance | Baseline and 12 months
  Short Physical Performance Battery (SPPB) will be used to evaluate this outcome. We will examine whether the exercise intervention alters SPPB performance.
Change in cognitively engaging activities | Baseline, 6 months and 12 months
  The Florida Cognitive Activity Scale (FCAS) will examine whether the exercise intervention altered engagement in cognitively stimulating activities or whether any outcomes varied as a function of cognitively stimulating activities. Scale 0-100, higher values = performing more cognitive stimulating activities.
Change in functional fitness | Baseline and 12 months
  Senior Fitness Test will be used to measure various aspects of fitness - e.g., balance, flexibility, strength. We will examine whether the exercise intervention improves any marker of fitness.
Incremental cost per quality adjusted life year (QALY) gained from the intervention | Baseline, 6 months, and 12 months
  Health resource utilization and quality of life measures will be used to calculate the costs per quality of adjusted life years. We will examine whether the intervention altered this metric.
Incremental Cost Effectiveness Ratio (ICER) | Baseline, 6 months, and 12 months
  Health resource utilization and quality of life measures will be used to calculate the costs per quality of adjusted life years. We will examine whether the intervention altered this metric.
Change in cortisol Levels | Baseline and 12 months
  Hair samples will be used to examine whether the exercise intervention altered hair cortisol, a measure of accumulated cortisol over several months.
Change in perceived cognitive abilities | Baseline and 12 months
  PROMIS Applied Cognition: (Abilities) This is a brief self-report of perceived cognitive abilities for daily functioning. We will examine whether the intervention alters this subjective/perceived level of cognitive function. Scale 8 -40, assess ppt. perceived functional abilities in regard to cognitive tasks. Higher value = higher self-perceived ability in cognition.
Gait speed | Baseline and 12 Months
  We will examine whether the intervention alters measures of gait speed under both single task and dual-task conditions.
Gait variability | Baseline and 12 Months
  We will examine whether the intervention alters measures of gait variability under both single task and dual-task conditions.
Change in Brain GSH levels | Baseline and 12 months
  MRI will be used to measure GSH levels. We will examine whether the exercise intervention alters levels of GSH.
History of Menopause and symptoms | Baseline
  Only given to female study participants. This questionnaire asks a variety of questions to gather information as it relates to menopause. We will examine whether any marker of neurocognitive performance or change in performance from the intervention varies in relation to reproductive history. We expect this to be used as a moderator in IGNITE. There is no scoring from this form, only recording in a yes:no fashion as to whether something happened or not. The frequency of any event will be examined as an effect moderator of the intervention.
Change in perceived concerns with cognition | Baseline and 12 months
  PROMIS Applied Cognition: (General Concerns) This is a brief self-report of perceived difficulties with cognition for daily functioning. We will examine whether the intervention alters this subjective/perceived level of cognitive function. Scale 8 -40. Lower score = less cognitive concerns
Change in level of daily functioning | Baseline and 12 month
  Everyday Cognition (ECOG)(Short version) measures subjective cognitive performance. We will examine whether the intervention alters this subjective/perceived level of cognitive function. Score range is 1 - 4 with lower scores equal to better daily function.
Change in exercise habits | Baseline and 12 months
  Godlin Leisure Time Exercise questionnaire is used to ask participants about usual leisure-time exercise habits. We will examine whether the intervention alters time spent in leisure time activities. Calculation of weekly minutes of activity into activity score, higher the score is equivalent to more active.
Current health status level | Baseline
  Cumulative Illness Rating Scale (CIRS): This scale is used to indicate the health status of older adults. Clinicians rate the pathology and impairment of major organ systems and also psychological, metabolic, neurological and musculoskeletal aspects of the individual. The CIRS consists of 14 aspects of health which are rated from 0 (no impairment to that organ/ system) to 4 (impairment is life threatening). We will examine whether the effectiveness of the intervention varies based on the comorbidity of various health conditions. Score range is 0-56 with lower score reflecting better health.
Change in levels of inactivity | Baseline, 6 months and 12 months
  Sitting Time Questionnaire scores how much time is spent sitting during 5 different events on a weekday and weekend day. We will examine whether participating in the intervention alters amount of time spent sitting. Calculate weekly minutes with higher values in minutes = more sedentary (sitting time)
Change in Self Esteem #1 | Baseline, 6 months and 12 months
  Self Esteem (PSPP): A 30-item instrument used to assess self-esteem relative to several domains of physical functioning in a hierarchical, multidimensional fashion. The instrument contains a general physical self-worth scale (PSW) which subsumes four more specific scales of perceived sport competence (SPORT), physical condition (COND), attractive body (BODY), and strength (STRENGTH), with six items per scale. Participants indicated on a four-point scale the degree to which each item is characteristic or true of them. Responses range from 1 (not at all true) to 4 (completely true).We will examine whether participating in the intervention alters measures of self-esteem. 4 subscales with score range 6 -24, higher number reflects more self esteem.
Change in Self Esteem #2 | Baseline, 6 months and 12 months
  Rosenberg Self-Esteem Scale (RSE): Widely-used scale in several domains of self- esteem research including physical activity. We will examine whether participating in the intervention alters measures of self-esteem. Scale 10 -50, higher values = higher levels of self esteem
Social support for study goal | Baseline and 12 Month
  Social Goal Importance: Asks the participant to name a friend, then rate how much that person helps or harms their pursuit of a personal goal. For this study, the goal in question is exercising/fitness. We will examine whether social goal importance relates to adherence to the intervention. Higher scores reflect more social support for the goals and lower scores reflect less social support for maintaining the goals.
Social Provisions | Baseline and 12 Month
  Social Provisions Scale (SPS):A 24-item scale assessing six relational provisions: attachment, or emotional support; social integration, or network support; reassurance of worth, or esteem support; reliable alliance, or tangible aid; guidance, or informational support; and the opportunity of nurturance.The items were modified for the exercise setting. For example, one of the statements used to assess social integration was "I feel part of the exercise group". We will examine whether social provisions relates to adherence to the intervention. Each subscale has range of 4 - 16 with total score range 24 - 96, higher values = higher social relationship (ppt. is receiving that provision)
Social Networks | Baseline and 12 Month
  Cohens Social Network Index: Self-report assessing the nature, quantity, and frequency of participants' social relationships. We will examine whether social provisions relates to adherence to the intervention or any of the neurocognitive outcomes. High contact in social networks have 0-12 score with higher number reflective of more social networks.
Relationship with exercise group/leader | Baseline, 6 Months and 12 Month
  Exercise Group Social Provisions Scale (EXSPS): 24 items related to the relationship between themselves and their exercise group/leader. Asks participants to rate on a scale of 1-4, with 1 being "strongly disagree" and 4 being "strongly agree." We will examine whether the relationship with the trainer influences adherence and compliance to the intervention. Score range 4 -16
Change in Healthy Eating Index (HEI) | Baseline and 12 Months
  Calculated via NCI Dietary (DHQ2). We will examine whether dietary habits moderate neurocognitive or physiological outcomes or change over the course of the intervention. Score range is 0-100 with higher numbers showing meeting key dietary recommendations and patterns.
Change in barriers to exercise | Baseline, 6 months and 12 months
  BARSE questionnaire assess degrees of confidence that one could exercise despite a variety of limitations such as during bad weather, while on vacation, etc. This scale was designed to tap subjects' perceived capabilities to exercise three times per week for 40 minutes over the next two months in the face of commonly identified barriers to participation. We will examine whether measures of barriers predicts adherence and compliance to the intervention. Scale 1-100, higher values = higher level of perceived capability to overcome barriers to exercise
Change in Glycemic Index (GI) | Baseline and 12 Months
  Calculated via NCI Dietary (DHQ2). We will examine whether the intervention alters measures of the glycemic index. It's a standardized score, range is -1 to 1. High scores mean that individuals consume a lot of the food items with high positive loading scores on the figure and low scores mean that people eat a low amount of food items with high positive loading scores (also likely more of the foods with negative loadings).
Change in Lifestyle Self Efficacy | Baseline, 6 months and 12 months
  Lifestyle Self-Efficacy (LSE): A 6-item measure to assess an individual's beliefs in their ability to accumulate 30 minutes of physical activity on 5 or more days of the week in the future. For each item, participants indicate their confidence to execute the behavior on a 100- point percentage scale comprised of 10-point increments, ranging from 0% (not at all confident) to 100% (highly confident). We will examine whether measures of self-efficacy predicts adherence and compliance to the intervention. Scale 0 -100, higher values = increased confidence to exercise 5 or more days per week for 30 minutes
Change in Exercise Self Efficacy | Baseline, 6 months and 12 months
  Exercise Self-Efficacy (EXSE): A 6-item measure to assess degrees of confidence in one's ability to continue exercising at moderate intensities 3 times per week for at least 40 minutes per session. We will examine whether measures of self-efficacy predicts adherence and compliance to the intervention. Scale 0 -100, higher values = higher confidence to continue to exercise (3X's week for 40 + minutes) in the future 8 weeks
Change in Self Regulation | Baseline, 6 months and 12 months
  Physical Activity Self-Regulation Scale, 12-item version (PASR-12): (PASR-12 FORM) A 12-item version of a popular 43-item self-regulation scale. Participants were asked to rate how often they used each strategy on a scale from 1 (never) to 5 (very often). We will examine whether measures of self-regulation predicts adherence and compliance to the intervention. Each subscale has range of 2 - 10, higher scores = greater use of self-regulation strategies. Summary score has range of 12 - 60
Change in Blood Pressure | Baseline and 12 months
  Measured as part of Pulse Wave Analysis. We will examine whether the intervention altered measures of blood pressure and whether these changes mediate neurocognitive changes.
Change in Oxygen Uptake Efficiency Slope (OUES) | Baseline and 12 months
  We will calculate this measure from the maximal exercise test and determine whether the exercise intervention improves OUES.
Exercise Adherence Volume | 12 months
  Study Participant level of adherence to prescribed volume of exercise minutes. We will examine how our intervention related to adherence (minutes per week) and whether better adherence relates to better cognitive outcomes.
Exercise Adherence Intensity | 12 months
  Study Participant level of adherence to prescribed intensity of exercise. We will examine how our intervention related to adherence (intensity zone) and whether better adherence relates to better cognitive outcomes.
Change in arterial stiffness | Baseline and 12 months
  This is measured by Carotid-Femoral Pulse Wave Velocity. This outcome is measured by capturing pulse pressure waveforms from the right carotid and femoral arteries using tonometry after 10 minutes of supine rest. We will examine whether the exercise intervention modified measures of arterial stiffness and how this relates to our various neurocognitive and physiological measures.
Fat mass | Baseline and 12 Months
  This will be assessed using a dual-energy x-ray absorptiometer (DXA). The DXA will provide a measure of fat mass from a total body scan. We will examine whether the exercise intervention alters measures of fat mass.
Change is waist circumference | Baseline and 12 Months
  The measurement will be completed at the midpoint between the lower rib and top of the iliac crest (hip bone) at the mid-axillary line. We will examine whether the exercise intervention alters measures of waist circumference.
Change in bone density | Baseline and 12 Months
  This will be assessed using a dual-energy x-ray absorptiometer (DXA). The DXA will provide a measure of Bone Density from a total body scan. We will examine whether the exercise intervention alters measures of bone density.

CONTACTS AND LOCATIONS:
Overall Officials: Kirk I Erickson, PhD, Principal Investigator — University of Pittsburgh
Locations (5):
- United States (5):
  - University of Illinois, Champaign, Illinois
  - University of Kansas, Kansas City, Kansas
  - Northeastern University, Boston, Massachusetts
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Carnegie Mellon University, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The data from this study will be made available to outside investigators under a data-sharing agreement. The data will be available to outside investigators after publication of the primary aims and at completion of quality control assessments and data organization. The investigators expect that the data from this study will result in significant interest from internal and external investigators for secondary data analysis and ancillary project proposals, so the investigators will create an oversight committee made up of Principal and Co-Investigators for monitoring, approving, and disseminating the data along with monitoring data analysis plans and development of manuscripts. This is important for eliminating redundant analyses, results, or manuscripts.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Will be made available after study investigators have published summary data and primary aim results. Will be available for unlimited amount of time.
Access Criteria: Data requests will be approved by IGNITE Executive committee. Requests can be made by completing data request form

REFERENCES:
- [Derived] Collins AM, Mellow ML, Wan L, Smith AE, Oberlin LE, Sewell KR, Gothe NP, Fanning J, Migueles JH, Dumuid D, Miatke A, Jakicic JM, Kang C, Grove G, Huang H, Sutton BP, Marsland AL, Kamboh MI, Kramer AF, Hillman CH, Vidoni ED, Burns JM, McAuley E, Erickson KI. Association between 24-h time-use composition and brain age: The IGNITE study. Alzheimers Dement (N Y). 2025 Dec 22;11(4):e70187. doi: 10.1002/trc2.70187. eCollection 2025 Oct-Dec. PMID 41445670
- [Derived] Norling AM, Lipsitz LA, Dufour AB, Travison TG, Sewell KR, Collins AM, Wan L, Grove G, Huang H, Oberlin LE, Jain S, Karikari TK, Morris JK, Jakicic JM, McAuley E, Kramer AF, Hillman CH, Vidoni ED, Billinger SA, Burns JM, Marsland AL, Kang C, Erickson KI. Arterial stiffness moderates the link between NfL and cognition: The IGNITE study. Alzheimers Dement. 2025 Aug;21(8):e70554. doi: 10.1002/alz.70554. PMID 40775489
- [Derived] Ripperger HS, Reed RG, Kang C, Lesnovskaya A, Aghjayan SL, Huang H, Wan L, Sutton BP, Oberlin L, Collins AM, Burns JM, Vidoni ED, Kramer AF, McAuley E, Hillman CH, Grove GA, Jakicic JM, Erickson KI. Cardiorespiratory fitness, hippocampal subfield morphology, and episodic memory in older adults. Front Aging Neurosci. 2024 Dec 19;16:1466328. doi: 10.3389/fnagi.2024.1466328. eCollection 2024. PMID 39749255
- [Derived] Raine LB, Erickson KI, Grove G, Watrous JNH, McDonald K, Kang C, Jakicic JM, Forman DE, Kramer AF, Burns JM, Vidoni ED, McAuley E, Hillman CH. Cardiorespiratory fitness levels and body mass index of pre-adolescent children and older adults during the COVID-19 pandemic. Front Public Health. 2023 Jan 17;10:1052389. doi: 10.3389/fpubh.2022.1052389. eCollection 2022. PMID 36733279

DOCUMENTS (1):
  • Informed Consent Form (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT02875301/ICF_000.pdf